CLINICAL TRIAL: NCT01364116
Title: The Accuracy of Noninvasive and Continuous Hemoglobin Measurement by Pulse CO-Oximetry™ in Children Undergoing Volume Expansion
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, assistant professor, Seoul National University Hospital
Other Study IDs: H-1012-127-346
Record Dates: First submitted 2011-05-24; First posted 2011-06-02 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Continuous Hemoglobin Measurement
Keywords: Pulse CO-Oximetry™; children; noninvasive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Measuring total hemoglobin(tHb) is a precious step to decide to start or to stop transfusion during operation. The newly developed instrument pulse CO-Cooximetry (Masimo) makes noninvasive monitoring of venous hemoglobin level (SpHb).

The objective of this study

* to compare the simultaneous level of tHb and SpHb during operation and after volume expansion in children
* to assess the accuracy of amount of acute change of SpHb on Masimo and tHb

ELIGIBILITY:
Inclusion Criteria: children under 10 years old how are diagnosed as

* brain tumor
* intraabdominal tumor
* intrathoracic tumor
* craniosynostosis
* scoliosis

Exclusion Criteria:

* cardiopulmonary disease
* preoperative infection
* genetic disease
* hematologic disease

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under 10 years old who were planned to take elective surgery which may cause patients' hemodynamic unstability.
  Patients who require intraoperative invasive arterial blood pressure monitoring.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-02; Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
hemoglobin concentrations from laboratory lab and pulse Co-oximetry | before and after volume expansion (20 minutes)
  volume expansion will be performed for 20 minuntes

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea